CLINICAL TRIAL: NCT00348816
Title: A Phase II Study to Assess the Feasibility and Activity of Concomitant Radiation and Docetaxel Chemotherapy Followed by Docetaxel Chemotherapy in Prostate Cancer Patients With a Persistent or Rising PSA After Radical Prostatectomy
Brief Title: Docetaxel, Radiation Therapy, and Prednisone in Treating Patients Who Have Undergone Surgery For Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000486733; HSC20050377H. (Other: UTHSCSA IRB)
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Prednisone; Radiotherapy

ARMS (1):
- Docetaxel (Single Arm) (Experimental): Docetaxel 20mg/m2/week IV every week during radiation treatment (7 cycles). Prednisone 5mg twice a day Radical prostatectomy as standard of care Radiation therapy will be used as standard of care Post radiation Doxcetaxel
  Interventions: Drug: docetaxel; Drug: prednisone; Procedure: Radical prostatectomy; Radiation: Radiation therapy

INTERVENTIONS:
Drug: docetaxel — Docetaxel 20mg/m2/week IV every week during standard of care radiation treatment (7 cycles). Post radiation: docetaxel 75mg/m2 IV every 21 days for 4 cycles plus prednisone 5mg PO BID QD.
  Other Names: Taxotere
Drug: prednisone — Docetaxel 20mg/m2/week IV every week during radiation treatment (7 cycles). Post radiation: docetaxel 75mg/m2 IV every 21 days for 4 cycles plus prednisone 5mg PO BID QD.
  Other Names: prednisone oral
Procedure: Radical prostatectomy — Radical prostatectomy as part of standard care
Radiation: Radiation therapy — Doses for standard care radiation therapy: The initial target volume will be the lower pelvis followed by a boost to the prostate fossa and immediate periprostatic tissue. The initial dose will be 4500 cGy. With the final boost, the total dose will be 6840-6900 cGy. (4500/25 plus 2340/13 or 2400/12) with a total of 37 or 38 fractions.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Docetaxel may make tumor cells more sensitive to radiation therapy. Giving docetaxel together with radiation therapy and prednisone after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving docetaxel together with radiation therapy and prednisone works in treating patients who have undergone surgery for prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the rate of prostate-specific antigen (PSA) decline and the number of patients reaching a PSA nadir of zero after treatment with chemoradiotherapy comprising docetaxel and external-beam radiotherapy followed by docetaxel and prednisone in patients with hormone-naive prostate cancer who have a persistent or rising PSA after radical prostatectomy.

Secondary

* Determine the tolerability of this regimen in these patients.
* Determine the progression-free survival, based on PSA progression, of these patients.
* Determine the overall survival of patients treated with chemoradiotherapy for rising PSA after radical prostatectomy.
* Determine if the velocity of subsequent PSA failure impacts survival of these patients.

Tertiary

* Document subsequent therapy for patients whose previous treatment has failed and if there is a response to that therapy.

Quaternary: To collect data on a contemporary cohort to those on study that received radiation alone. We will match cancer and patient characteristics to determine if the variable of chemotherapy has any impact on outcomes.

OUTLINE: Patients receive docetaxel IV over 1 hour on days 1, 8, 15, 22, 29, 36, and 43 and undergo external-beam radiotherapy on days 1-5, 8-12, 15-19, 22-26, 29-33, 36-40, and 43-47.

Beginning within 6 weeks after completion of chemoradiotherapy, patients receive docetaxel IV over 1 hour on day 1 and oral prednisone twice daily on days 1-21. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 1 month, every 4 months for 2 years, and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer
* Prostate-specific antigen (PSA) level > 0.2 ng/mL after radical prostatectomy performed ≥ 6 weeks ago
* No lymph node-positive prostate cancer
* No documented metastatic disease

  * CT scan of the abdomen and pelvis negative (within the past 6 months)
  * No bone pain OR negative bone scan (within the past 6 months)
* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Bilirubin normal
* ALT and AST ≤ 1.5 times upper limit of normal
* Alkaline phosphatase normal
* Fertile patients must use effective contraception
* No peripheral neuropathy > grade 1
* No other malignancy within the last 5 years that could affect the diagnosis or assessment of prostate cancer
* No serious illness with a life expectancy of < 5 years
* No concurrent medical, psychological, or social circumstance that would preclude study compliance
* No history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80

Exclusion Criteria:

* No prior orchiectomy
* No prior chemotherapy regimen for this disease
* No prior pelvic radiotherapy
* No pre- or postoperative androgen manipulation, such as luteinizing hormone-releasing hormone agonists, antiandrogens (flutamide, bicalutamide, or nilutamide), or finasteride

  * Preoperative androgen manipulation for a duration of ≤ 3 months allowed
* No prior immunotherapy
* No prior strontium chloride Sr 89, samarium Sm 153 lexidronam pentasodium, or other systemic radioisotopes
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)
* No concurrent herbal or alternative regimens including, but not limited to, any of the following:

  * Saw palmetto
  * PC-SPES
  * Shark cartilage
* No other concurrent investigational agents
* No other concurrent chemotherapy, immunotherapy, or hormonal therapy (except for replacement steroids)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-05; Primary Completion 2016-07-08 (Actual); Study Completion 2016-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory P. Swanson, MD, Study Chair — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment opened on 21 Mar 2006 and closed on 15 Apr 2009. The first subject was consented on 18 May 2007 and the final subject on 14 Apr 2009. Subjects were all enrolled in outpatient clinics and received treatment as outpatients.
Pre-assignment Details: Subjects must have histologic diagnosis of prostate cancer and be post prostatectomy. They must have a PSA > 0.2 ng/ml (verified on 2 separate tests, at least 2 weeks apart). CT abdomen/pelvis and bone scan must be negative. One subject was a screen failure due to CT showed lung mass (not related to prostate cancer).
Groups:
- Docetaxel (Single Arm): Docetaxel 20mg/m2/week IV every week during radiation treatment (7 cycles). Post radiation: docetaxel 75mg/m2 IV every 21 days for 4 cycles plus prednisone 5mg PO BID QD.
  Adjuvant therapy: radical prostatectomy as part of standard care
  Radiation therapy: Doses for standard care radiation therapy: The initial target volume will be the lower pelvis followed by a boost to the prostate fossa and immediate periprostatic tissue. The initial dose will be 4500 cGy. With the final boost, the total dose will be 6840-6900 cGy. (4500/25 plus 2340/13 or 2400/12) with a total of 37 or 38 fractions.
Period: Overall Study
Arm/Group | Docetaxel (Single Arm)
Started | 20
Completed | 19
Not Completed | 1
Not completed — Noncompliance with radiation treatment | 1

BASELINE CHARACTERISTICS:
Population: 21 patients were consented, 1 patient was screen failure due to lung mass found during staging.
Arm/Group | Docetaxel (Single Arm)
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 65 [48 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Rate of Prostate-Specific Antigen (PSA) Decline Reported as the Number of Subjects Reaching a PSA Nadir of Zero Following the Intervention.
Description: Subjects were followed after the intervention and monitored for PSA (Prostate Specific Antigen) decline for up to 5 years of follow-up, to determine how many had a decline and reached a PSA nadir of zero..
Time Frame: 5 years
Population: Exceptions to group description: (1) one subject non-compliant and taken off study (not included in analysis); (2) one subject did not receive docetaxel #7 during radiation due to change in performance status; (3) one subject received only 1 post radiation docetaxel; (4) two subjects did not receive post radiation docetaxel #4.
Measure: Count of Participants; unit: Participants
Groups:
- Docetaxel (Single Arm): Docetaxel 20mg/m2/week IV every week during radiation treatment (7 cycles). Post radiation: docetaxel 75mg/m2 IV every 21 days for 4 cycles plus prednisone 5mg PO BID QD. Doses for standard care radiation therapy: The initial target volume will be the lower pelvis followed by a boost to the prostate fossa and immediate periprostatic tissue. The initial dose will be 4500 cGy. With the final boost, the total dose will be 6840-6900 cGy. (4500/25 plus 2340/13 or 2400/12) with a total of 37 or 38 fractions.
Arm/Group | Docetaxel (Single Arm)
Number analyzed (Participants) | 19
Participants | 12

2. Secondary Outcome: Progression-free Survival Based on PSA Progression
Description: Subjects were monitored for PSA (Prostate Specific Antigen) for up to 5 years of follow-up.
Time Frame: 5 years
Population: One subject was not included in analysis due to taken off study due to non-compliance
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel (Single Arm)
Number analyzed (Participants) | 19
Participants | 12

3. Secondary Outcome: Overall Survival
Time Frame: 5 years
Population: N/A no data recorded
Groups:
- Overall Survival: N/A, no data for overall survival recorded
Arm/Group | Overall Survival
Number analyzed (Participants) | 0

4. Secondary Outcome: Correlation Between Velocity of Subsequent PSA Failure and Survival
Time Frame: 5 years
Population: N/A no study data was recorded for this outcome
Groups:
- Correlation Between Velocity of Subsequent PSA Failure and Sur: All study completers
Arm/Group | Correlation Between Velocity of Subsequent PSA Failure and Sur
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From time of consent to 5 years post treatment.
Arm/Group | Docetaxel (Single Arm)
All-Cause Mortality (participants affected / at risk) | 12/20
Serious Adverse Events (participants affected / at risk) | 12/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel (Single Arm) (N=20)
Infection - other: (Infections and infestations) | 1 (3) — URI, Lung (pneumonia), Pleura (empyema)
Febrile neutropenia (Infections and infestations) | 1 (1)
Stricture/Stenosis GU: Bladder Neck (Renal and urinary disorders) | 2 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 3 (3) — Thigh abscess, port, uroma
Pain - Other: Cardiac (Cardiac disorders) | 2 (2)
Colitis Infectious (Infections and infestations) | 1 (1) — Clostridium difficile
Cardiac General - Other: (Cardiac disorders) | 2 (2) — Cardiac Artery Bypass
Allergic Reaction (Immune system disorders) | 1 (1) — Lisinopril
CNS cerebrovascular ischemia (Nervous system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Musculoskeletal/Soft Tissue - Other: total knee arthroplasty (Musculoskeletal and connective tissue disorders) | 1 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Left femoral head
Mood alteration (Psychiatric disorders) | 2 (3) — Bipolar, off medication (hospitalized twice) and anxiety attack
Dizziness (Nervous system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 1 (1) — Subdural
Renal Failure (Renal and urinary disorders) | 1 (1)
Renal/Genitourinary-Other: Artificial Urinary Sphincter (Renal and urinary disorders) | 1 (1)
Renal/Genitourinary-Other: Removal of foreign body (Renal and urinary disorders) | 1 (1) — Surgery clips
Urinary retention (Renal and urinary disorders) | 1 (4)
Dehydration (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel (Single Arm) (N=20)
Allergic reaction (Immune system disorders) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 18 (18)
Anorexia (Gastrointestinal disorders) | 1 (1)
Blurred vision (Eye disorders) | 3 (3)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (2)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cystitis (Renal and urinary disorders) | 9 (12)
Diarrhea (Gastrointestinal disorders) | 18 (26)
Dizziness (Nervous system disorders) | 7 (8)
Dry eye symdrome (Eye disorders) | 1 (1)
Dry mouth/salivary gland (xerotomia) (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dermatology/Skin-Other: Boil on back, I&D no growth (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin-Other: Rash with pruritus (Skin and subcutaneous tissue disorders) | 1 (1) — Preexisting on arms, legs and back that worsened during treatment
Dermatology/Skin-Other: seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Erectile dysfuncion (Reproductive system and breast disorders) | 5 (5)
Edema: head and neck (General disorders) | 3 (3)
Edema: limb (General disorders) | 4 (4)
Fatigue (General disorders) | 16 (26)
Flu-like syndrome (General disorders) | 10 (12)
Gastrointestinal, other: teeth grinding (Gastrointestinal disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (8)
Gynecomastia (Reproductive system and breast disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 4 (4)
Hemoglobin (Blood and lymphatic system disorders) | 14 (34)
Hemorrhage, GI: rectum (Gastrointestinal disorders) | 11 (12)
Hemorrhage, GU: Urinary NOS (Renal and urinary disorders) | 5 (5)
Hemorrhage, pulmonary/upper respiratory: nose (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hot flashes (Endocrine disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (episode after infusion) (Vascular disorders) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 11 (13)
Infection, other: URI (Infections and infestations) | 4 (4)
Infection, other: tooth (Infections and infestations) | 1 (1)
Infection, other: urinary (Infections and infestations) | 1 (2)
Infection, other: perineal (Infections and infestations) | 1 (1)
Infection with normal ANC (port)(UTI)(balanitis-penis) (Infections and infestations) | 5 (6)
Insomnia (Psychiatric disorders) | 11 (12)
Joint and/or muscle pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Leukocytes (total WBC) (Investigations) | 8 (35)
Libido (Psychiatric disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 7 (7)
Mood alteration (anxiety, emotion, irritability, depression, mood swings) (Psychiatric disorders) | 6 (7)
Mucositis/stomatitis (Gastrointestinal disorders) | 2 (2)
Nail changes (Skin and subcutaneous tissue disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 8 (12)
Neuropathy: Motor (Nervous system disorders) | 1 (1)
Neuropathy: Sensory (Nervous system disorders) | 15 (16)
Neurology, other: Dementia (Nervous system disorders) | 1 (1)
Neutrophiles/granulocytes (ANC/AGC) (Investigations) | 5 (16)
Ocular/Visual-Other: light sensitivity (Eye disorders) | 1 (1)
Otitis (non-infectious) (Ear and labyrinth disorders) | 1 (1)
Pain: Back (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain: Breast (Reproductive system and breast disorders) | 1 (1)
Pain: Cardiac/heart (Cardiac disorders) | 2 (2)
Pain: Extremity/limb (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain: Headache (Nervous system disorders) | 6 (6)
Pain: Oral cavity (gum soreness under dentures) (Gastrointestinal disorders) | 1 (1)
Pain: Perineum (Gastrointestinal disorders) | 1 (1)
Pain: Port (Surgical and medical procedures) | 1 (1)
Pain: Scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Pain: Scrotum (Reproductive system and breast disorders) | 2 (2)
Pain: Shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain: Teeth (Gastrointestinal disorders) | 2 (4)
Pain: Throat (Gastrointestinal disorders) | 1 (1)
Pain: Urination (Renal and urinary disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 16 (17)
Pulmonary/Upper Respiratory, other: Viral bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary/Upper Respiratory, other: sinus fullness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash: dermatitis associated with radiation (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 6 (6)
Rigors/Chills (General disorders) | 1 (1)
Sexual/Reproductive Function-Other: Erection, involunary, painful) (Reproductive system and breast disorders) | 1 (1)
Stricture/stenosis GU: bladder neck (Renal and urinary disorders) | 3 (3)
Stricture/stenosis GU: urethra (Renal and urinary disorders) | 2 (2)
Supraventricular and nodal arrhythmia: tachycardia (Cardiac disorders) | 1 (1)
Taste alteration (Gastrointestinal disorders) | 9 (9)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Urinary frequency/urgency (Renal and urinary disorders) | 9 (13)
Urinary retention (Renal and urinary disorders) | 1 (7)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Viral hepatitis (Infections and infestations) | 1 (1)
Vision-flashing lights/floaters (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes